CLINICAL TRIAL: NCT05265325
Title: A Phase 2, Multicenter, Open-label, Randomized, Active-Controlled Study of Efficacy and Safety of AND017 in the Treatment of Anemia in Patients With Chronic Kidney Disease on Dialysis
Brief Title: A Study of AND017 to Treat Anemia in Chronic Kidney Disease Patients on Dialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kind Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AND017-MN-202
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Renal Anemia
MeSH Terms: interventions — Epoetin Alfa; Darbepoetin alfa; continuous erythropoietin receptor activator

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- AND017 Dose Regimen A (Experimental): AND017 will be administrated orally at dose A three times a week
  Interventions: Drug: AND017 capsules TIW
- AND017 Dose Regimen B (Experimental): AND017 will be administrated orally at dose B once a week
  Interventions: Drug: AND017 capsules QW
- Erythropoietin stimulating agent (Active Comparator): Investigator will select an erythropoietin stimulating agent, such as epoetin alfa, darbepoetin alfa, Mircera®, or their biosimilars, for the patient under this arm with starting doses and dose adjustment rules according to the epoetin alfa USPI or SmPC.
  Interventions: Drug: epoetin alfa, darbepoetin alfa, Mircera®, or their biosimilars

INTERVENTIONS:
Drug: AND017 capsules TIW — Orally, 3 times per week in Period 1 and dose adjustment in Period 2 at 2 mg/4 mg and 2-weeks interval according to Hb levels
  Arms: AND017 Dose Regimen A
Drug: AND017 capsules QW — Orally, once per week in Period 1 and dose adjustment in Period 2 at 4 mg/8 mg and 2-weeks interval according to Hb levels
  Arms: AND017 Dose Regimen B
Drug: epoetin alfa, darbepoetin alfa, Mircera®, or their biosimilars — Dose regimen and adjustment rules according to the USPI or SmPC or local practice
  Arms: Erythropoietin stimulating agent

SUMMARY:
This is a phase II study to evaluate the safety and efficacy of AND017 in renal anemia patients on dialysis

DETAILED DESCRIPTION:
This is a Phase II study to assess the safety and efficacy of AND017 in patients with CKD who are anemic and on dialysis.

ELIGIBILITY:
Key Inclusion Criteria:

1. Body weight from 45 to 140 kg inclusive
2. Receiving stable HD (including combination methods such as hemodiafiltration or hemofiltration), HHD, or PD for ESKD for a minimum of 16 weeks prior to randomization and determined by the Investigator to be compliant with dialysis treatment prescription.
3. Patient must have been on IV or SC of an approved ESA under the prescription for at least 6 weeks, and ≤25% change in dose between the two most recent doses, prior to randomization.
4. The mean of two hemoglobin values during screening (at least 7 days apart) must be 9.0-11.0 g/dL with a difference of ≤1.3 g/dL between the two values
5. TSAT ≥ 20% or ferritin ≥ 100 ng/mL at screening
6. Folate ≥ 3.0 ng/mL and vitamin B12 ≥ lower limit of normal (LLN) at screening
7. AST and ALT < 3×ULN at screening.
8. No evidence of other causes of anemia caused by a pathologic process in the hematopoietic system, including intra- or extravascular hemolysis, or myelodysplasia.

Key Exclusion Criteria:

1. Concurrent retinal neovascular lesions requiring treatment including proliferative diabetic retinopathy, exudative age-related macular degeneration, retinal vein occlusion, macular edema, etc.
2. Anemia determined by the Investigator to be caused by concurrent autoimmune disease with inflammatory symptoms (such as systemic erythematosus, ankylosing spondylitis, rheumatoid arthritis, psoriatic arthritis, Sjögren's syndrome, celiac disease, etc.).
3. History of gastric/intestinal resection considered influential on the absorption of drugs in the gastrointestinal tract (excluding resection of gastric or colon polyps) or concurrent symptomatic gastroparesis despite on treatment.
4. Clinically significant bleeding (eg, requiring transfusion or drop in Hb of ≥ 2 g/dL) within 4 weeks of first dose; bleeding diathesis or risk of bleeding that has not been medically or surgically corrected at least 4 weeks prior to first dose of study drug.
5. Uncontrolled hypertension defined as patients with hypertension having more than one of three diastolic blood pressure values >95 mmHg and each test at least 5 min apart during the screening assessment.
6. Concurrent congestive heart failure (New York Heart Association [NYHA] Class III or higher).
7. History of stroke, transient ischemic attack (TIA), myocardial infarction, thromboembolic event (deep vein thrombosis, DVT), pulmonary embolism, or lung infarction within 24 weeks before the screening assessment.
8. Positive for hepatitis B surface antigen or anti-hepatitis C virus antibody at the screening assessment, or positive for human immunodeficiency virus in a past test.
9. Not complying with COVID-19 prevention and control requirements per local policy.
10. Concurrent primary form of anemia other than renal anemia (hemolytic anemia, thalassemia, sickle cell anemia, history of pure red cell aplasia, history of myelodysplastic syndrome or multiple myeloma, iron deficiency, etc.). Any question of the primary cause of anemia should be discussed with the Medical Monitor before the patient signs informed consent.
11. Known hemosiderosis, hemochromatosis or hyper-coagulable condition
12. Known to be hypersensitive or intolerant to ESA.
13. Having received treatment with androgenic anabolic steroids, testosterone enanthate, or mepitiostane within 5 weeks prior to the first dose.
14. Any treatment with a hypoxia-inducible factor prolyl hydroxylase inhibitor (HIF-PHI) within 5 weeks prior to the first dose.
15. TBIL>1.5 ULN, or AST>3 ULN, or ALT>3 ULN, or ALP>3 ULN, or previous or concurrent serious liver disease (acute or active chronic hepatitis, cirrhosis, etc.) thought to be caused by any other HIF-PHI.
16. Previous or current malignant tumor (patients with no recurrence for at least 5 years are eligible. Exemption: basal cell and squamous cell carcinoma not under active stage).
17. Patients with a history of significant liver disease or active liver disease.
18. Patients that have major surgery planned during the study period.
19. Patients that have undergone blood transfusion or with evidence of major blood loss within 8 weeks before the screening assessment. Investigators should discuss this with the Medical Monitor for cases where there is doubt about whether to exclude or not.
20. Patients unable to discontinue IV iron during the screening period.
21. Patients with an organ transplant on immunosuppression, or with a scheduled kidney or any other organ transplant within the duration of the study, or without kidney.
22. Serum albumin < 2.5 g/dL at screening.
23. Patients with other chronic medical condition that may limit life expectancy in the opinion of the Investigator.
24. History of a seizure disorder or any occurrence of seizures in the past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 20 weeks
  Incidence of adverse events
Mean change from baseline in Hb at Week 6 | Up to 5 weeks after dosing
  Mean change from baseline in Hb at Week 6

SECONDARY OUTCOMES:
Proportion of responders, during the entire study period. | up to Week 20
  Responders are defined as patients whose Hb achieved ≥ 10.0 g/dL and an increase ≥ 1.0 g/dL from baseline
Mean proportion of visits at which patients maintain Hb within the target range from baseline during the fixed-dose period and titration period | up to Week 20
  Target range is defined as 10.0-11.0 g/dL inclusive and an increase ≥ 1.0 g/dL.
Proportion of patients with a mean Hb between 10.0-11.0 g/dL inclusive during Week 14-20 | at Week 14, 15, 16, 17, 18, 19, and 20
  Proportion of patients with a mean Hb between 10.0-11.0 g/dL inclusive during Week 14-20
Change in Hb from baseline to the mean Hb levels over Week 14-20 | Baseline and at Week 14, 15, 16, 17, 18, 19, and 20
  Change in Hb from baseline to the mean Hb levels over Week 14-20
Mean Hb levels and mean change from baseline in Hb level at each visit | up to Week 20
  Mean Hb levels and mean change from baseline in Hb level at each visit
Cumulative response rate over the entire study period | up to Week 20
  Response is defined as Hb < 10.0 g/dL or an increase in hemoglobin of <1 g/dL from baseline

OTHER OUTCOMES:
EPO levels and change from baseline at each visit | up to Week 20
  EPO levels and change from baseline at each visit
Hepcidin levels and change from baseline at each visit | up to Week 20
  Hepcidin levels and change from baseline at each visit
Iron study levels and change from baseline at each visit | up to Week 20
  Iron study levels and change from baseline at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Yusha Zhu, MD, PhD, Study Director — Kind Pharmaceuticals LLC
Locations (25):
- United States (10):
  - US Renal Care - Pine Bluff, Pine Bluff, Arkansas
  - North America Research Institute, Riverside, California
  - Rocky Mountain Kidney Care, Lone Tree, Colorado
  - Nephrology and Hypertension Specialists, Dalton, Georgia
  - High Desert Nephrology Associates, Gallup, New Mexico
  - Nephrology Associates of Western New York, Cheektowaga, New York
  - Nephrology Consultants of Northwest Ohio - Toledo, Toledo, Ohio
  - South Texas Renal Care Group - San Saba, San Antonio, Texas
  - Clinical Advancement Center PLLC, San Antonio, Texas
  - South Texas Renal Care Group, San Antonio, Texas
- China (15):
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Xiamen Branch, Zhongshan hospital affilicated to Fudan University, Xiamen, Fujian
  - Xiamen Fifth Hospital, Xiamen, Fujian
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hunan
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - Zhongshan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Jinshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Zigong First People's Hospital, Zigong, Sichuan